CLINICAL TRIAL: NCT01710670
Title: A Double-blind, Randomized, Placebo-controlled, Three-way Crossover Study to Investigate the Drug-Drug Interactions of Brivaracetam and Ethanol in Healthy Male Subjects.
Brief Title: A Study to Investigate the Drug-Drug Interactions of Brivaracetam and Ethanol in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EP0041; 2012-002591-14 (EudraCT Number)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2012-12

CONDITIONS: Healthy Volunteers
Keywords: Brivaracetam; Ethanol; Pharmacodynamics; Pharmacokinetic; Interaction
MeSH Terms: interventions — brivaracetam; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ethanol + Brivaracetam (Experimental): Treatment A: Ethanol + Brivaracetam
  Interventions: Drug: Brivaracetam; Other: Ethanol
- Ethanol Placebo + Brivaracetam (Experimental): Treatment B: Ethanol Placebo + Brivaracetam
  Interventions: Drug: Brivaracetam; Other: Ethanol Placebo
- Ethanol + Brivaracetam Placebo (Experimental): Treatment C: Ethanol + Brivaracetam Placebo
  Interventions: Other: Ethanol; Other: Brivaracetam Placebo

INTERVENTIONS:
Drug: Brivaracetam — Strength: 200 mg (4 x 50 mg)
  Form: oral tablet
  Frequency: single dose
  Description: All subjects will receive a single oral dose of Brivaracetam (BRV) 200 mg, given as 50 mg tablets times 4 followed by an adequate volume of water (approximately 200 ml) in 2 of the 3 crossover periods. This dose will be administered 30 minutes after the initiation of the Ethanol / Ethanol Placebo infusion on Day 1.
  Arms: Ethanol + Brivaracetam; Ethanol Placebo + Brivaracetam
Other: Ethanol — Form: intravenous infusion
  Frequency: continuous infusion
  Description: The ethanol infusion rate is initially based on weight, height, age, and sex. Subsequently, the infusion rate will be adjusted based on Breath Ethanol Measurements to maintain Breath Ethanol Levels (and by extension, blood ethanol levels) of 0.6 g / L.
  Arms: Ethanol + Brivaracetam; Ethanol + Brivaracetam Placebo
Other: Brivaracetam Placebo — In 1 of the 3 crossover periods, all subjects will receive 4 Placebo tablets to match the 50 mg Brivaracetam (BRV) tablets. The Placebo tablet will contain the same excipients as the BRV tablets but without BRV.
  Arms: Ethanol + Brivaracetam Placebo
Other: Ethanol Placebo — In 1 crossover period subjects will receive Ethanol Placebo (5% glucose). On Day 1, the continuous infusion of Ethanol Placebo will begin with a 30 minute Loading Phase prior to administration of Brivaracetam (BRV) / BRV Placebo and will continue until 5 hours after administration of BRV/BRV Placebo. During the first 10 minutes, the infusion will be accompanied by an infusion of 5% Glucose via the same line in order to mask the sensation at the beginning of the Ethanol infusion.
  Arms: Ethanol Placebo + Brivaracetam

SUMMARY:
To evaluate if Brivaracetam (BRV) influences the psychomotor and cognitive impairing effects of Ethanol

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers with the age between 18 and 55 years old

Exclusion Criteria:

* Subject has participated or is participating in any other clinical studies of investigational drug or another investigational medical product within the last 3 months or has participated in 4 or more Investigational Medicinal Product (IMP) studies within 1 year prior to screening
* Subject is not healthy (eg, taking any drug treatments except use of Paracetamol, excessive amount of alcohol, cigarettes, caffeine consumption, having a positive drug / alcohol abuse, having abnormal safety parameters)
* Subject has not been vaccinated for hepatitis
* Subjects has consumed any grapefruits, grapefruits juice, grapefruit-containing products or star fruit within 14 days prior to dosing or not able to refrain from these products during the study
* Subject has Ethanol intolerance
* Subject has a known hypersensitivity to any components of the Investigational Medicinal Product (IMP)
* Subject has made a blood donation or a comparable blood loss (500 ml) within the last 3 months prior to screening
* subject is an employee of the investigator or study center or subject is a first line family member of an employee working in the respective study center or of the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Saccadic Eye Movements from 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  Average values of Latency (reaction time), Saccadic Peak Velocity, and Inaccuracy (difference between stimulus angle and corresponding saccade in percentages) will be calculated for all artifact-free saccades.
Smooth pursuit eye movements from 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  The time during which the eyes are in smooth pursuit of the target will be calculated for each frequency and expressed as a percentage of stimulus duration. The average percentage of smooth pursuit for all stimulus frequencies will be used as a parameter.
Adaptive tracking from 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  Performance will be scored after a fixed period of 3.5 minutes and reflected visuo motor control and vigilance. The average performance scores will be used in the analysis.
Body sway from 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  The body sway meter allows measurement of body movements in a single plane, providing a measure of postural stability. (antero-posterior sway in mm / 2 minutes)
Visual Analog Scales for Mood From 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  Visual Analog Scales according to Bond and Lader
Visual Analog Scale for alcohol intoxication From 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  The scale consists of a 10 cm line anchored on the left end by "sober" and on the right end by "drunk." Subjects mark a point on the line that best represents their subjective state corresponding to the condition tested. The result is a distance calculated from the mark on the line.
Visual Verbal Learning Test from 1.5 hours Post-Dose up to 6 hours Post-Dose | From 1.5 hours Post-Dose up to 6 hours Post-Dose
  Immediate recall, immediate recognition, delayed recall, and delayed recognition to evaluate memory
Visual Analog Scales for Alertness From 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  Visual Analog Scales according to Bond and Lader
Visual Analog Scales for Calmness From 60 minutes Pre-Dose up to 10 hours Post-Dose | From 60 minutes Pre-Dose up to 10 hours Post-Dose
  Visual Analog Scales according to Bond and Lader

SECONDARY OUTCOMES:
The area under the plasma concentration-time curve from zero to infinity (AUC) | From Pre-Dose (- 5 minutes) to 36 hours Post-Dose
  Blood samples will be taken - 5 minutes Pre-Dose, 15, 30, and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours Post-Dose.
The area under the plasma concentration-time curve from zero to the time of the last measured concentration above the limit of quantification [AUC(0-t)] | From Pre-Dose (- 5 minutes) to 36 hours Post-Dose
  Blood samples will be taken - 5 minutes Pre-Dose, 15, 30, and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours Post-Dose.
The maximum plasma concentration (Cmax) | From Pre-Dose (- 5 minutes) to 36 hours Post-Dose
  Blood samples will be taken - 5 minutes Pre-Dose, 15, 30, and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours Post-Dose.
The time to reach the maximum plasma concentration (tmax) | From Pre-Dose (- 5 minutes) to 36 hours Post-Dose
  Blood samples will be taken - 5 minutes Pre-Dose, 15, 30, and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours Post-Dose.
The terminal disposition rate constant (λz) with the respective terminal half-life (t1/2) | From Pre-Dose (- 5 minutes) to 36 hours Post-Dose
  Blood samples will be taken - 5 minutes Pre-Dose, 15, 30, and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours Post-Dose.
Serum Ethanol concentrations | From - 30 minutes Pre-Dose to 10 hours Post-Dose
  Blood samples for Ethanol concentrations will be taken - 30 minutes, - 15 and - 5 minutes Pre-Dose, then 15, 30 and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, and 10 hours Post-Dose.
Breath Ethanol concentrations | From - 30 minutes Pre-Dose to 10 hours Post-Dose
  Blood samples for Ethanol concentrations will be taken - 30 minutes, - 15 and - 5 minutes Pre-Dose, then 15, 30 and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, and 10 hours Post-Dose.
Total Ethanol Dose analyzed by a model independent parameter estimate | From - 30 minutes Pre-Dose to 10 hours Post-Dose
  Blood samples for Ethanol concentrations will be taken - 30 minutes, - 15 and - 5 minutes Pre-Dose, then 15, 30 and 60 minutes Post-Dose and then 2, 3, 4, 5, 6, 8, and 10 hours Post-Dose.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Leiden, Netherlands